CLINICAL TRIAL: NCT04501770
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity Profiles of the Recombinant Anti-HER2 and Anti-CD3 Humanized Bispecific Antibody (M802) in HER2-Positive Advanced Solid Tumors
Brief Title: A Study of M802 (HER2 and CD3) in HER2-Positive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M80201
Record Dates: First submitted 2020-07-31; First posted 2020-08-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: HER2-Positive Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M802 (Experimental): Subjects who meet the enrollment criteria will enter the core treatment period and receive a cycle of treatment with M802 (once weekly for 4 weeks) via intravenous infusion. And eligible subjects who complete the core treatment period will receive a cycle of extended treatment (once weekly for 4 weeks) until disease progression or toxicity intolerance.
  Interventions: Drug: Chort 1 of M802; Drug: Chort 2 of M802; Drug: Cohort 3 of M802; Drug: Cohort 4 of M802; Drug: Cohort 5 of M802; Drug: Cohort 6 of M802; Drug: Cohort 7 of M802; Drug: Cohort 8 of M802

INTERVENTIONS:
Drug: Chort 1 of M802 — Cohort 1, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 2 μg, and the maintenance dose during core treatment period and extended treatment period is 5 μg.
Drug: Chort 2 of M802 — Cohort 2, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 5 μg, and the maintenance dose during core treatment period and extended treatment period is 10 μg.
Drug: Cohort 3 of M802 — Cohort 3, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 10 μg, and the maintenance dose during core treatment period and extended treatment period is 20 μg.
Drug: Cohort 4 of M802 — Cohort 4, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 20 μg, and the maintenance dose during core treatment period and extended treatment period is 50 μg.
Drug: Cohort 5 of M802 — Cohort 5, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 50 μg, and the maintenance dose during core treatment period and extended treatment period is 100 μg.
Drug: Cohort 6 of M802 — Cohort 6, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 100 μg, and the maintenance dose during core treatment period and extended treatment period is 150 μg.
Drug: Cohort 7 of M802 — Cohort 7, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. Dose on D1 is 150 μg, and on D8, D15, D22 is 225 μg.
Drug: Cohort 8 of M802 — Cohort 8, subjects will be administered M802 via intravenous infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. The starting dose is 225 μg, and the maintenance dose during core treatment period and extended treatment period is 300 μg.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of different doses of M802 in patients with HER2-positive advanced solid tumors, and to determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) so as to provide basis for the recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥18 years old.
2. Patients must have a diagnosis of histologically or cytologically confirmed metastatic advanced solid tumor with failure to standard treatment and who have no available therapy that may confer clinical benefit. Patients with HER2-positive metastatic breast cancer should have received standard anti-HER2 therapies.
3. HER2 expression status report should be provided during the screening period with fluorescence in-situ hybridization (FISH) or Chromogenic in situ hybridization (CISH) test positive, or immunohistochemistry IHC 3+, or immunohistochemistry IHC 2+ and confirmed by amplification of FISH or CISH.
4. Patients must have stopped anti-tumor treatment for at least 4 weeks prior to the first dose of M802. The anti-tumor treatment includes chemotherapy, immunotherapy, targeted therapy, endocrine therapy, and radiotherapy (except for local radiation therapy for alleviating pain, at least 14 days after end of treatment).
5. Patients must have measurable lesions at baseline according to the RECIST Version 1.1.
6. Patients must have an ECOG performance status (PS) Score of 0-1.
7. Patients must have an expected survival > 12 weeks.
8. Patients must have a baseline left ventricular ejection fraction (LVEF) ≥ 50%.
9. Patients must have adequate haematological and organ functions as indicated by the following laboratory values:

   Haematological: Absolute Neutrophil Count (ANC) ≥ 1.5 ×10^9/L; Blood Platelet Count (BPC) ≥ 80 ×10^9/L; Hemoglobin ≥ 9.0 g/dL (No blood transfusions within 14 days).

   Hepatic: Bilirubin ≤ 1.5 × upper limit of normal (ULN); AST and ALT ≤ 2.5 × ULN (AST, ALT ≤ 5 × ULN is allowed when there is liver metastasis).

   Renal: Serum creatinine ≤ 1.5 × ULN.
10. Patients must understand and voluntarily agree to participate by signing written informed consent.

Exclusion Criteria:

1. Patients who had prior treatment with trastuzumab or similar monoclonal drugs within 4 weeks before first dosing of M802.
2. Patients with brain metastasis.
3. Patients who have uncontrollable active infections (Grade ≥ 2 according to CTCAE Version 5.0).
4. Patients with severe respiratory disease who are not suitable for the study at the judgment of investigator.
5. Patients with severe immunosuppression (long-term use of immunosuppressant or glucocorticoid with daily dosage of dexamethasone ≥10 mg).
6. Patients who have other malignant tumors in the past 5 years, except the complete cured cervical carcinoma in situ or basal cell or squamous cell carcinoma.
7. Patients with a history of serious cardiovascular disease, including receiving coronary artery bypass grafts or coronary stenting, occurrence of myocardial infarction, congestive heart failure within 6 months, or a history of unstable angina, uncontrolled severe hypertension or arrhythmia requiring medication.
8. Patients with a history of autoimmune diseases (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
9. Patients with severe hyperthyroidism or hypothyroidism.
10. Patients with metabolic diseases such as uncontrolled diabetes, severe gastrointestinal bleeding, severe diarrhea (Grade ≥ 2 according to CTCAE Version 5.0), or severe gastrointestinal obstruction requiring intervention.
11. Patients with a history of immunodeficiency, including HIV positive.
12. Patients with Hepatitis b surface antigen test positive or hepatitis c antibody test positive.
13. Patients who have received inoculation of (attenuated) live virus vaccine within 4 weeks before first dosing of M802.
14. Pregnant, lactating women, or females or males who have fertility plan within 12 months.
15. Patients with a previous history of definite neurological or psychiatric disorders, including epilepsy or dementia.
16. Patients who participated in clinical studies of other drugs within 4 weeks prior to first dosing of M802 (using last dosing of other drug's clinical studies as end).
17. Patients with adverse reactions from previous treatment haven't recovered to grade 1 according to CTCAE Version 5.0 (except for residual effect on hair loss).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
MTD | From the time of first dosing (Day 1) until the forth dosing (Day 28)
  Number of DLTs (dose limiting toxicities) during the first 28 days after the first administrations of study drug in each cohort.
RP2D | From the start of administration to the end of the study or 28 days after the administration is stopped (up to 1 years and 28 days)
  Incidence and severity of AEs, and SAEs, including but not limited to laboratory values, PK and biomarkers. All AEs will be classified as Grades 1 through 5 as defined by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Area under the curve (AUC) of M802 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The endpoints for assessment of PK of M802 include serum concentrations of M802 at different timepoints after M802 administration.
Maximum observed concentration (Cmax) of M802 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The endpoints for assessment of PK of M802 include serum concentrations of M802 at different timepoints after M802 administration.
Minimum observed concentration (Cmin) of M802 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The endpoints for assessment of PK of M802 include serum concentrations of M802 at different timepoints after M802 administration.
Expression levels of CEA | From the time of screening period until disease progression or toxicity intolerance (up to 1 years and 28 days).
  As tumor marker, expression levels of CEA will be tested in hospitals.
Expression levels of CA15-3 | From the time of screening period until disease progression or toxicity intolerance (up to 1 years and 28 days).
  As tumor marker, expression levels of CA15-3 will be tested in hospitals.
Expression levels of CA125 | From the time of screening period until disease progression or toxicity intolerance (up to 1 years and 28 days).
  As tumor marker, expression levels of CA125 will be tested in hospitals.
Expression levels of CA19-9 | From the time of screening period until disease progression or toxicity intolerance (up to 1 years and 28 days).
  As tumor marker, expression levels of CA19-9 will be tested in hospitals.
Expression levels of CA72-4 | From the time of screening period until disease progression or toxicity intolerance (up to 1 years and 28 days).
  As tumor marker, expression levels of CA72-4 will be tested in hospitals.
Cytokines | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The levels of pharmacodynamic cytokines will be determined at the PD central laboratory.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The immunogenicity of M802 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
The antibody titer of the neutralizing antibody | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  The immunogenicity of M802 will be collected by testing the antibody titer of the neutralizing antibody.
ORR | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  Objective response rate (ORR) is defined as the proportion of patients with complete response (CR) and partial response (PR), based on RECIST Version 1.1.
DCR | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 1 years).
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response (CR) and partial response (PR), based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- wuhan YZY Biopharma Co.,Ltd., Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No